CLINICAL TRIAL: NCT01483859
Title: Prediction of Intraoperative Blood Loss and Postoperative Recovery by Liver Stiffness Measurement (Fibroscan®) in Right Hepatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Jeong-Rim LEE, Assistant Professor, Yonsei University
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 1-2011-0053
Record Dates: First submitted 2011-11-24; First posted 2011-12-01 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-07

CONDITIONS: Liver Malignancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- right hepatectomy with preoperative LSM (Other): patients undergoing right hepatectomy with preoperative LSM between August 2007 and July 2011
  Interventions: Other: preoperative liver stiffness measurement

INTERVENTIONS:
Other: preoperative liver stiffness measurement — Liver stiffness measurement (LSM) using Fibroscan is a newly introduced noninvasive tool that generates an elastic wave using a vibrator applied to the thoracic wall at the level of the right lobe of the liver and measures the prolongation velocity of the wave, which is directly associated with liver stiffness (LS).
  Other Names: Liver stiffness measurement (LSM) using Fibroscan®(EchoSens, Paris, France)

SUMMARY:
Liver stiffness measurement (LSM) using Fibroscan®(EchoSens, Paris, France) is a newly introduced noninvasive tool that generates an elastic wave using a vibrator applied to the thoracic wall at the level of the right lobe of the liver and measures the prolongation velocity of the wave, which is directly associated with liver stiffness (LS). Although recent advances in surgical techniques and perioperative management have made with established perioperative management have now made it possible to perform hepatectomies as a safe procedure with minimum mortality, the possibility of massive blood loss and resultant transfusion during hepatectomy still exist. The objective of this research was to identify the role of liver stiffness measurement for the prediction of intraoperative blood loss and postoperative recovery after elective right hepatectomy.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing right hepatectomy between August 2007 and July 2011

Exclusion Criteria:

* patients undergoing right hepatectomy without preoperative liver stiffness measurement

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-09; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The correlation between the value of liver stiffness measurement and intraoperative blood loss during right hepatectomy | Participants will be followed for perioperative period, approximate 6 weeks through chart review.
  The investigators will investigate the value of liver stiffness measurement and intraoperative blood loss during right hepatectomy through chart review. The investigators will analyze the correlation between the value of liver stiffness measurement and intraoperative blood loss during right hepatectomy

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Severance Hospital, Seoul, Seoul
  - Severance Hospital, Seoul